CLINICAL TRIAL: NCT01604551
Title: Membrane Shedding During Severe Sepsis and Septic Shock: Pathophysiological and Clinical Relevance
Brief Title: Membrane Shedding During Septic Shock
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 4649
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2012-05

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Microparticles (MPs) result from plasma cell membrane remodeling and shedding after cell stimulation or apoptosis. MPs are know recognized as a pool of bioactive messengers with emerging role in pathophysiology of immune and cardiovascular diseases. MPs have been characterized during septic shock and may contribute to dissemination of pro-inflammatory and procoagulant mediators. This is a prospective observational study of circulating MPs and blood coagulation in 100 septic shock patients admitted in 3 tertiary hospitals medical ICU at baseline (D1), D2, D3, D4 and D7.

ELIGIBILITY:
Inclusion Criteria:

* Septic shock
* Informed consent

Exclusion Criteria:

* Class IV heart failure
* Child-Plugh grade C cirrhosis
* Cancer under active treatment
* BMI>35 kg/m²
* Moribund patient
* DNR decision

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with septic shock
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2003-05; Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xavier DELABRANCHE, MD, Principal Investigator — Service de Réanimation Médicale, Nouvel Hôpital Civil, Hôpitaux Universitaires de Strasbourg, France
Locations (3):
- France (3):
  - Service Réanimation Médicale et Médecine Hyperbare, CHU, Angers
  - Centre Hospitalier, Mulhouse
  - Service de Réanimation Médicale, Nouvel Hôpital Civil, Hôpitaux Universitaires, Strasbourg